CLINICAL TRIAL: NCT06199076
Title: Experimental Study on Alcohol Use and Behavior in Young Adults
Acronym: OXYCAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Halted due to recruitment problems.
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Joar Guterstam, PhD, M.D., Psychiatrist, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-501809-13-01
Record Dates: First submitted 2023-12-13; First posted 2024-01-10 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Oxytocin/Placebo, Alcohol Use Disorder (Experimental): Visit 1: Alcohol Use Disorder participants will receive 24 IU of oxytocin prior to completing behavioral task measures
  Visit 2: Alcohol Use Disorder participants will receive 24 IU of placebo (saline solution) prior to completing behavioral task measures
  Interventions: Drug: Oxytocin nasal spray
- Placebo/Oxytocin, Alcohol Use Disorder (Experimental): Visit 1: Alcohol Use Disorder participants will receive 24 IU of placebo (saline solution) prior to completing behavioral task measures
  Visit 2: Alcohol Use Disorder participants will receive 24 IU of oxytocin prior to completing behavioral task measures
  Interventions: Drug: Oxytocin nasal spray
- Oxytocin/Placebo, Healthy Control (Experimental): Visit 1: Healthy Control participants will receive 24 IU of oxytocin prior to completing behavioral task measures
  Visit 2: Healthy Control participants will receive 24 IU of placebo (saline solution) prior to completing behavioral task measures
  Interventions: Drug: Oxytocin nasal spray
- Placebo/Oxytocin, Healthy Control (Experimental): Visit 1: Healthy Control participants will receive 24 IU of placebo (saline solution) prior to completing behavioral task measures
  Visit 2: Healthy Control participants will receive 24 IU of oxytocin prior to completing behavioral task measures
  Interventions: Drug: Oxytocin nasal spray

INTERVENTIONS:
Drug: Oxytocin nasal spray — The clinical trial is a phase II-study double-blind placebo-controlled study. The trial will have a parallel group cross-over design where subjects with alcohol use disorder versus healthy controls will administer a single dose of intranasal oxytocin versus placebo on two study visits 1-3 weeks apart.
  Other Names: Syntocinon Intranasal Spray

SUMMARY:
The goal of this double blind randomized placebo-controlled clinical trial is to compare intranasal oxytocin and placebo in young adult individuals with alcohol use disorder as compared to healthy controls. The main questions it aims to answer are:

* The effect of oxytocin versus placebo on prosocial behavior in individuals with high- versus low alcohol use
* The effect of oxytocin versus placebo on impulsivity, emotion recognition, social learning, and alcohol craving in individuals with high- versus low alcohol use

Participants in both groups will on two separate visits perform the following validated behavioral task measures:

* Dictator game tasks assessing prosocial behavior
* Delay discounting task assessing impulsivity
* Emotion recognition task assessing emotion recognition
* Alcohol cue craving task assessing alcohol craving
* Observational fear learning task assessing social learning

Researchers will compare groups of high and low alcohol use to see if there is a difference in effect of oxytocin versus placebo between groups.

DETAILED DESCRIPTION:
Hypotheses:

1. OXT vs. placebo will improve the deficits in prosocial behavior in individuals with AUD vs. HC,
2. OXT vs. placebo will improve the deficits in impulsivity, difficulties in emotion recognition and social learning in AUD vs. HC
3. OXT vs. placebo will reduce craving for alcohol, in individuals AUD vs. HC

Material and Methods:

The study will include young adults (18-24 years old): 110 individuals with AUD and 110 healthy controls (HC) matched on gender, education, and age. Sample size estimation is based on effect sizes from previous studies investigating prosocial behavior in addiction, and studies on the influence of OXT on social cognition respectively.

Both groups will undergo thorough psychiatric assessment before inclusion and eligible participants will be invited to a two-session laboratory study (2 weeks apart) randomized for the order of administration of the study compound. On the planned test day after controlling for alcohol and drug use, intranasal OXT and matching placebo at a dose of 24IU will be administered. Behavioral tasks previously developed in our laboratory and evaluated in AUD populations to identify social cognitive impairments in terms of prosocial behavior and emotion recognition will be utilized. In addition, validated behavioral measure of impulsivity, namely the Delay discounting task will be used and craving will be assessed by a standardized assessment battery developed by our laboratory which includes a combination of a standardized questionnaire and visual cues comprising images of alcohol and people drinking.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years of age
* Male
* Give informed consent and comply with study procedure
* Understands written Swedish

Alcohol use disorder (AUD) group

* Fulfils criteria for at least moderate AUD the past 12 months according to MINI Neuropsychiatric Interview
* Fulfils at least 8 points on the Alcohol Use Disorder Identification Test

Healthy control group

* No criteria for AUD the past 12 months according to MINI Neuropsychiatric Interview
* Fulfils less than 8 points on the Alcohol Use Disorder Identification Test

Exclusion Criteria:

* Fulfils criteria for any substance use disorder (except AUD for AUD-group, and mild cannabis- and nicotine use disorder for both groups).
* Using cocaine, amphetamines, hallucinogens, benzodiazepines, etc. within 1 month of the start of the study (excluding cannabis)
* Cannabis use more than 2 days in past month
* Cannabis use on day of testing or day before testing
* Traces of alcohol as measured by breathalyzer on the day of testing
* History of severe psychiatric disorder (e.g. severe depression, bipolar, antisocial personality disorder) or neuropsychiatric disorder of ADHD, autism or Tourette's.
* Medical conditions of such severity that they require continual clinical attention, such as regular follow-up visits, prescribed medications or other specific treatment
* Prescription medicine the past 3 months
* Using non-prescription medicine that could not be stopped 48 hours prior to each visit
* Using intranasal medicine that could not be stopped 48 hours prior to each visit
* Prescription medicine the past 3 months
* Allergy or intolerance to preservatives in nasal spray, e.g. latex allergy.
* Upper-respiratory tract infection (i.e. a 'common cold' resulting in significant nasal congestion) at day of testing (but with the possibility of rescheduling for another time point)
* History of nasal disease (e.g. atrophic rhinitis, recurrent nose bleeds), nose damage (e.g. broken nose), and nasal surgery
* History of head trauma (i.e. loss of consciousness longer than 2 minutes)
* Simultaneous participation in another clinical trial

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-representation, i.e., sex assigned as male at birth.
Enrollment: 206 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Prosocial behavior using a brief 2-trial dictator game task measured at both study visits. | 35-45 minutes after administration of the investigational medicinal product
  Prosocial behavior using a Dictator game task previously developed and evaluated for a alcohol use disorder population. Subjects are informed that they will be anonymous and play online with other anonymous interaction partners. The subject is asked to decide and indicate their distribution of points for oneself and/or another subject. Prosocial behavior will be operationalized as the points transferred to the other subjects on each trial. Time approx: 5 minutes.
Prosocial behavior using an extended dictator game task measured at both study visits. | 46-65 minutes after administration of the investigational medicinal product
  Prosocial behavior using a Dictator game task previously developed and evaluated for assessing the effect of oxytocin on prosocial behavior. Subjects are informed that they will be anonymous and play online with other anonymous interaction partners. The subject is asked to decide and indicate their preference regarding the distribution of points for oneself and/or another subject. Prosocial behavior will be operationalized as the proportional preference of self/other point distribution. Time approx: 15 minutes.

SECONDARY OUTCOMES:
Impulsivity using a delay discounting task task measured at both study visits. | 76-80 minutes after administration of the investigational medicinal product.
  The subject decides on whether to keep a smaller number of points today, or a larger number of points in the future operationalized as the discounting rate. Time approx: 5 minutes.
Emotion recognition using an emotion recognition task measured at both study visits. | 81-90 minutes after administration of the investigational medicinal product.
  The subject identifies the correct emotion from a set facial expression images. Time approx: 10 minutes.
Alcohol craving using an alcohol cue-craving task measured at both study visits. | 91-110 minutes after administration of the investigational medicinal product.
  The subject is in separate steps presented with alcohol cues for their preferred beverage (e.g. beer or wine) with increasing intensity while alcohol craving being measured using the Alcohol Urge Questionnaire. Time approx: 10 minutes.
Social learning using an observational fear learning task measured at both study visits. | 111-120 minutes after administration of the investigational medicinal product.
  The subject observes a video of an allegedly previous subject receiving mild electric stimulation in conjunction to watching some colored squares on a screen while skin conductance is being measured. Time approx: 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Joar Guterstam, PhD, M.D., Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Division of Psychology, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No